CLINICAL TRIAL: NCT05665738
Title: Two-fraction High Dose Rate Brachytherapy as Monotherapy Delivered Three Hours Apart in Localized Prostate Cancer: A Pilot Study
Brief Title: Two-fraction HDR Monotherapy for Localized Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23721; NCI-2024-01993 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Prostate Adenocarcinoma; Localized Prostate Carcinoma
Keywords: Brachytherapy; Radiotherapy; High Dose Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- HDR brachytherapy (Experimental): Participants will receive the same radiotherapy technique, methods, and delivery will as standard of care 3 hours apart instead of receiving the radiotherapy on separate days.
  Interventions: Radiation: High Dose Rate Monotherapy

INTERVENTIONS:
Radiation: High Dose Rate Monotherapy — High dose rate brachytherapy delivered in 13.5 Gy x 2 fractions over a single implant procedure 3 hours apart
  Other Names: HDR Monotherapy; High dose rate brachytherapy

SUMMARY:
This is a single center single arm prospective pilot study investigating the safety of high dose rate (HDR) brachytherapy as monotherapy delivered in 2 fractions 3 hours apart. HDR monotherapy has been established as safe and effective in this context, however previous studies have delivered 2 fractions on separate days, or at least 6 hours apart. Clinically, this regimen, if shown to be safe and effective in future studies, has the potential to reduce operative resources and logistical stresses on brachytherapy departments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of HDR monotherapy 13.5 Gy x 2 fractions delivered 3 hours apart in patients with low and intermediate risk prostate cancer.

SECONDARY OBJECTIVES:

I. To describe the prostate specific antigen (PSA) kinetics associated with HDR brachytherapy monotherapy 13.5 Gy x 2 fractions delivered 3 hours apart for low and intermediate risk prostate cancer.

OUTLINE:

Treatment will be administered on an outpatient basis. All treatment will be delivered over a single day. Participants will be followed for 6 months after last treatment or removal from study, or until death, whichever occurs first. Additional Follow up will be as per usual guidelines for prostate cancer, every 3 months following treatment with PSA for the first year, then every 4 months after year 2, and every 6 months after year 3 until 5 years of follow up are completed.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically or cytologically confirmed diagnosis of prostate adenocarcinoma.
2. National Comprehensive Cancer Network low to intermediate risk stratification.
3. No prior treatment for prostate cancer and no prior androgen deprivation therapy.
4. Age >=18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status <2 (Karnofsky >60%.
6. Eligible to undergo High dose rate (HDR) brachytherapy as monotherapy as determined by the treating radiation oncologist.
7. Ability to understand and the willingness to sign a written informed consent document.
8. Human immunodeficiency virus (HIV)-infected individuals on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
9. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
10. Individuals with a history of hepatitis C virus (HCV) infection must have been treated and cured. For individuals with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
11. Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria:

1. Any prior treatment for prostate cancer.
2. Any prior androgen deprivation therapy.
3. Is currently receiving any other investigational agents.
4. Abnormal pre-brachytherapy assessment raising concern for undergoing HDR brachytherapy procedure.
5. Contraindications to general anesthesia.
6. Contraindications to radiotherapy.
7. Prior cryosurgery or cryotherapy to the prostate.
8. Prior transurethral resection of the prostate within the previous 6 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with treatment-related adverse events | Up to 6 months
  The proportion of participants with reported grade 3 or higher genitourinary (GU) or gastrointestinal (GI) toxicities, as graded by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be reported.

SECONDARY OUTCOMES:
Mean Prostate Specific Antigen (PSA) Nadir | Up to 6 months
  The mean (average) PSA nadir after treatment will be reported along with standard deviations.
Mean Time to PSA Nadir | Up to 6 months
  The mean (average) time to PSA nadir after treatment will be reported along with standard deviations.
Mean Change in International Prostate Symptom Score (IPSS) over time | Up to 6 months
  The mean change over time on scores for the International Prostate Symptom Score (IPSS) will be reported along with standard deviations. The IPSS measures the severity of lower urinary tract symptoms and erectile function with lower numbers indicating less change in symptoms. Seven questions with scores ranging from 1-5 are summed to create a total score. Scores of 1-7 indicate mild symptoms, scores of 8-19 indicate moderate symptoms, and scores of 20-35 indicate severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: I-Chow Hsu, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martell K, Mendez LC, Chung HT, Tseng CL, Alayed Y, Cheung P, Liu S, Vesprini D, Chu W, Wronski M, Szumacher E, Ravi A, Loblaw A, Morton G. Results of 15 Gy HDR-BT boost plus EBRT in intermediate-risk prostate cancer: Analysis of over 500 patients. Radiother Oncol. 2019 Dec;141:149-155. doi: 10.1016/j.radonc.2019.08.017. Epub 2019 Sep 12. PMID 31522882
- [Background] Viani GA, Arruda CV, Assis Pellizzon AC, De Fendi LI. HDR brachytherapy as monotherapy for prostate cancer: A systematic review with meta-analysis. Brachytherapy. 2021 Mar-Apr;20(2):307-314. doi: 10.1016/j.brachy.2020.10.009. Epub 2021 Jan 15. PMID 33461894
- [Background] Morton G, McGuffin M, Chung HT, Tseng CL, Helou J, Ravi A, Cheung P, Szumacher E, Liu S, Chu W, Zhang L, Mamedov A, Loblaw A. Prostate high dose-rate brachytherapy as monotherapy for low and intermediate risk prostate cancer: Efficacy results from a randomized phase II clinical trial of one fraction of 19 Gy or two fractions of 13.5 Gy. Radiother Oncol. 2020 May;146:90-96. doi: 10.1016/j.radonc.2020.02.009. Epub 2020 Mar 5. PMID 32146259
- [Background] Alayed Y, Loblaw A, McGuffin M, Chung HT, Tseng CL, D'Alimonte L, Cheung P, Liu S, Chu W, Szumacher E, Helou J, Ravi A, Haider M, Mamedov A, Zhang L, Morton G. Single-fraction HDR brachytherapy as monotherapy in low and intermediate risk prostate cancer: Outcomes from two clinical trials with and without an MRI-guided boost. Radiother Oncol. 2021 Jan;154:29-35. doi: 10.1016/j.radonc.2020.09.007. Epub 2020 Sep 10. PMID 32918971
- [Background] Corkum MT, Achard V, Morton G, Zilli T. Ultrahypofractionated Radiotherapy for Localised Prostate Cancer: How Far Can We Go? Clin Oncol (R Coll Radiol). 2022 May;34(5):340-349. doi: 10.1016/j.clon.2021.12.006. Epub 2021 Dec 25. PMID 34961659
- [Background] Kukielka AM, Dabrowski T, Walasek T, Olchawa A, Kudzia R, Dybek D. High-dose-rate brachytherapy as a monotherapy for prostate cancer--Single-institution results of the extreme fractionation regimen. Brachytherapy. 2015 May-Jun;14(3):359-65. doi: 10.1016/j.brachy.2015.01.004. Epub 2015 Feb 28. PMID 25736733